CLINICAL TRIAL: NCT00958048
Title: Effects of Early Intervention With Nocturnal Non-invasive Ventilation in Patients With Amyotrophic Lateral Sclerosis: A Randomized, Controlled Trial
Brief Title: Effects of Nocturnal Non-invasive Ventilation in Patients With Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200812112R; 2011-04-011LA (Other: Taipei Veterans General Hospital)
Record Dates: First submitted 2009-02-08; First posted 2009-08-13 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2013-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; hypoventilation
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Hypoventilation | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Experimental): ALS with non-invasive ventilation
  Interventions: Device: non-invasive ventilation
- 1 (No Intervention): ALS without non-invasive ventilation

INTERVENTIONS:
Device: non-invasive ventilation — CPAP, BiPAP
  Arms: 2

SUMMARY:
Specific aims:

Aim 1. To determine the incidence of hypoventilation in Amyotrophic Lateral Sclerosis (ALS) patients.

Aim 2. To identify the clinical characteristics and risk factors associated .

Aim 3. To determine the effect of early intervention with nocturnal NIV on the prognosis of ALS patients.

DETAILED DESCRIPTION:
Objectives: Amyotrophic lateral sclerosis is the commonest motor neuron disease with incidence of 0.8 person-years in Chinese. Respiratory muscle function has been proposed to be a strong predictor of quality of life (QoL) and survival in ALS. Some studies suggest that most patients with ALS developed hypoventilation when their vital capacity (FVC) is less than 50% of predicted value. However, the incidence of hypoventilation and factors associated with hypoventilation in ALS patients is not clear. Also, there is still no consensus as to which physiologic marker should be used as a trigger for the initiation of non-invasive ventilation (NIV) in ALS patients. The conflicts of studies come from variable subgroup of ALS, pulmonary function at enrollment, techniques used to diagnose ALS, time to apply NIV, and target endpoint. Therefore, this project aimed to study ALS patients who had relatively preserved respiratory muscle function and no respiratory failure at clinical to achieve three goals: (1) To determine the incidence of hypoventilation in ALS patients (2) To identify the clinical characteristics and risk factors associated with hypoventilation in ALS patients (3) To determine the effect of early intervention with NIV on the prognosis of ALS patients Study design: Randomized, controlled trial Participants: ALS patients whose FVC 40%-80% of predict, Pimax <60mmHg, and daytime PaCO2<50mmHg Protocol: Eligible patients with whole-night polysomnography (PSG) and transcutaneous CO2 (PtcCO2). Enrolled patients were randomized to standard treatment or NIV. The primary endpoint of prognosis was survival. The secondary endpoint was changes of PtcCO2 and PaCO2, unexpected admission or clinic visiting, daytime function and QoL.

Statistic: The baseline demographics of patients with or without hypoventilation were compared to determine the factors associated with hypoventilation in ALS patients. The impact of NIV in ALS patients was determined by comparing the primary and secondary goals between standard treatment and NIV group. A two-sided p value of < 0.05 was considered statistically significant.

Clinical implication: Hypoventilation at ALS patients who had relatively preserved respiratory muscle function and no respiratory failure at clinical sleep was common, early identification through PSG screening and PtcCO2 will allow for the early diagnosis and intervention. Understanding the time of applying NIV and the effect on prognosis in ALS will allow for the early intervention and prediction of outcomes.

ELIGIBILITY:
Inclusion Criteria:

* ALS patients who:

  * had FVC 40%-80% of predict
  * Pimax < 60 mmHg
  * daytime PaCO2 < 50 mmHg

Exclusion Criteria:

* Refuse to participate
* Require mechanical ventilation
* Active neurologic event other than ALS
* Obstructive pulmonary disease
* Active infection
* Need sedatives or narcotics within 3 days of sleep study
* Participating in other study at the same time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Survival | 36 months

SECONDARY OUTCOMES:
Changes of PtcCO2 and PaCO2, admission or unexpected clinical visiting, and QoL | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Peilin Lee, M.D., Principal Investigator — National Taiwan University Hospital; Whey Dong Wu, M.D., Principal Investigator — Naitonal Taiwan University Hospital
Locations (1):
- Peilin Lee, Taipei, Taiwan